CLINICAL TRIAL: NCT02749045
Title: The Simultaneous Assessment of Invasive Fractional Flow Reserve and SPECT Myocardial Ischemia Using Regadenoson in the Catheterization Laboratory
Brief Title: Simultaneous Assessment of FFR and SPECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment, funding period ended
Sponsor: Prem Soman (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Prem Soman, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO15090404
Record Dates: First submitted 2016-03-03; First posted 2016-04-22 (Estimated); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Image acquisition arm (Other): Subjects who have undergone a clinically indicated fractional flow reserve measurement in the cardiac catheterization laboratory will receive standard dose Tc-99m sestamibi and undergo resting SPECT image acquisition within three hours from end of cardiac catheterization procedure.
  Interventions: Radiation: SPECT imaging

INTERVENTIONS:
Radiation: SPECT imaging — myocardial perfusion imaging

SUMMARY:
The overall purpose of this research study is to identify the disparity in ischemia measurement between fractional flow reserve (FFR) used in the cardiac catheterization laboratory and myocardial perfusion stress- single-photon emission computed tomography (SPECT). This study aims to determine the correlation between simultaneous FFR and SPECT obtained using regadenoson in the catheterization laboratory.

DETAILED DESCRIPTION:
Patients who are previously scheduled for diagnostic coronary angiography will be approached for consent to be part of the study. If the patient is found to have one or two vessel disease and it is planned by the interventional cardiologist that FFR will be used, then the previously consented patient will be deemed appropriate for the study. The standard procedure will be followed for FFR testing using regadenoson. The patient will then receive the standard dose of Tc-99m sestamibi. The interventional cardiologist will proceed with percutaneous coronary intervention (PCI) if appropriate. Patients will proceed to the cardiac catheterization laboratory holding area post procedure. Patients will then be scheduled to be taken to the nuclear cardiology laboratory one to three hours following the coronary angiogram for standard SPECT acquisition. Patients will be monitored for 2-6 hours or overnight as clinically indicated following diagnostic coronary angiography and PCI. Low dose resting myocardial perfusion scanning may be performed the next day if stress myocardial perfusion study was abnormal.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing clinically-indicated FFR measurement (to determine the hemodynamic significance of intermediate degrees of stenosis) for single or two -vessel epicardial coronary disease during diagnostic coronary angiography for suspected coronary artery disease.

Exclusion Criteria:

1. Patients with 3-vessel disease
2. Prior coronary artery bypass grafting
3. Patients with second or third- degree atrioventricular block, without a functioning pacemaker
4. Patients who have ingested caffeine-containing products within the past 12 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-07; Primary Completion 2020-12 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prem Soman, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was significantly affected by COVID-19 and the increasing use of iFR in place of FFR
Period: Overall Study
Arm/Group | Image Acquisition Arm
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Image Acquisition Arm
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Concordance Between Gated SPECT Perfusion Data (QGS) and Fractional Flow Reserve (FFR)
Description: The concordance will be calculated as the percentage of patients who had an abnormal FFR (<0.8) and an abnormal SPECT (a perfusion defect on the SPECT) PLUS patients who had a normal FFR (≥ 0.8) and a normal SPECT.
  concordance= patients with abnormal FFR and abnormal SPECT + patients with normal FFR and normal SPECT/ total no. of patients
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Image Acquisition Arm
Number analyzed (Participants) | 27
Participants | 19

ADVERSE EVENTS:
Time Frame: Adverse events related to Tc-99m sestamibi SPECT occurring during the patient's stay in the nuclear lab (3-4 hours) were recorded.
Arm/Group | Image Acquisition Arm
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

LIMITATIONS AND CAVEATS:
The study was significantly under-recruited. A pre-hoc power calculation indicated that a minimum of 50 patients was required to produce meaningful results. Recruitment was affected by: 1) the increasing use of iFR in place of FFR in the cath lab, and 2) COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02749045/Prot_SAP_000.pdf